CLINICAL TRIAL: NCT06943703
Title: Safety, Efficacy, and Long-Term Outcomes of Intralesional Bleomycin Injection as an Adjunctive Therapy for Pediatric Lymphatic Malformations: A Retrospective Study on Cosmetic and Health-Related Quality of Life Improvements.
Brief Title: Bleomycin as an Effective and Curative Adjunct Therapy for Lymphangioma
Status: Completed | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Nguyen Thanh Quang, Pediatric surgeon, National Children's Hospital, Vietnam
Other Study IDs: VUNI.2223.SG04
Record Dates: First submitted 2025-04-06; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Lymphangioma; Lymphatic Malformations
Keywords: Bleomycin; Lymphangioma; Lymphatic malformations; Intralesional Bleomycin injection; Sclerotherapy; Quality of life; Pediatric vascular anomalies; Head and neck; Safety and efficacy; Cosmetic; Non-surgical; Abdominal; Axilla; Thorax
MeSH Terms: conditions — Lymphangioma; Lymphatic Abnormalities | interventions — Sclerotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric Patients with Lymphangiomas Treated with Intralesional Bleomycin: This cohort consists of pediatric patients under the age of 18, diagnosed with lymphangiomas (lymphatic malformations), treated at the National Children's Hospital between 2018 and 2022. The lymphangiomas in this group are most commonly located in the head and neck, but may also occur, though less frequently, in the axilla, abdomen, thorax, groin, and extremities. The patients included in this cohort were selected based on their diagnosis of lymphangiomas without serious comorbidities that could complicate treatment or outcomes of the sclerotherapy. These patients were managed or observed during the study period, and the cohort represents a diverse age range of children under 18.
  Interventions: Drug: Sclerotherapy with intralesional bleomycin injection

INTERVENTIONS:
Drug: Sclerotherapy with intralesional bleomycin injection — The intervention studied is intralesional Bleomycin injection, which involves the direct injection of Bleomycin, a chemotherapeutic agent, into the lymphangioma lesions. This minimally invasive procedure is aimed at reducing the size of the lymphangioma by disrupting the abnormal growth of lymphatic vessels. The dosage of Bleomycin is tailored based on the patient's body weight, typically ranging from 1 to 3 mg per kg of body weight per injection. The intervention is distinct from other treatments, such as surgical excision or other sclerotherapy agents, as it specifically utilizes Bleomycin's mechanism of action to induce tissue sclerosis and promote lesion regression without the need for invasive surgery. This intervention may require multiple treatment sessions, depending on the size, location of the lymphangioma, and individual's response to therapy, with the goal of achieving long-term effectiveness and improving cosmetic outcomes.

SUMMARY:
Lymphatic malformations (LM), or lymphangiomas, are common vascular anomalies in children, most often occurring in the head and neck, less commonly in the axilla, abdomen, thorax, groin, and extremities. These benign but locally invasive lesions can cause complications such as respiratory issues, difficulty swallowing, nerve compression, bleeding, and cosmetic disfigurement. Treatment traditionally involves surgical excision, but this approach carries risks such as nerve damage, high recurrence, and poor cosmetic results. In recent years, sclerotherapy, specifically Bleomycin injection, has emerged as a less invasive alternative, offering potential benefits like reduced recurrence and better cosmetic outcomes.

Since its introduction in Vietnam in 2016, Bleomycin has been used to treat LM, but comprehensive studies on its safety, efficacy, and long-term outcomes in pediatric patients are lacking. This study aims to fill this gap by evaluating the effectiveness of intralesional Bleomycin injections in children with LM treated at the National Children's Hospital between 2018 and 2022.

The study will assess the safety, efficacy, and long-term outcomes of Bleomycin, focusing on lesion size reduction, recurrence rates, and cosmetic and health-related quality of life (QoL) improvements. The retrospective study will involve more than 800 pediatric patients and use tools like the Patient Scar Assessment Questionnaire (PSAQ) and Short Form-36 (SF-36) health survey to evaluate cosmetic outcomes and overall well-being.

The research will also compare the effectiveness of Bleomycin alone versus in combination with surgery, examining whether Bleomycin can reduce the need for additional interventions. By offering a comprehensive evaluation of both clinical and patient-reported outcomes, the study aims to establish Bleomycin as a viable, minimally invasive treatment option for pediatric LM, improving both clinical and cosmetic outcomes for these patients.

In addition, this study will provide valuable local data on Bleomycin's use in Vietnam, potentially influencing national treatment guidelines. The results will be disseminated in peer-reviewed journals, contributing to global understanding of Bleomycin's role in managing lymphatic malformations in children.

DETAILED DESCRIPTION:
Lymphatic malformations (LM), often referred to as lymphangiomas, are a form of vascular malformation that arises due to the abnormal development of the lymphatic system. These benign but locally invasive lesions are one of the most common vascular anomalies in children. The highest incidence of lymphangiomas is seen in the head and neck region, where they can cause a range of serious complications such as respiratory obstruction, dysphagia (difficulty swallowing), and nerve compression. Less commonly locations of lymphangiomas include axilla, abdomen, thorax, groin, and extremities which could cause bleeding, compression of adjacent structures, and visible deformity, pain and discomfort. Left untreated, these malformations can lead to significant morbidity and functional impairment, as well as severe cosmetic disfigurement, particularly in pediatric patients.

Historically, surgical excision has been the primary treatment for lymphangiomas. However, this approach carries several risks, including damage to surrounding vital structures such as nerves and blood vessels, high recurrence rates due to incomplete excision, and unsightly scars. Over the last few decades, sclerotherapy (ST) has emerged as a less invasive, more favorable alternative that reduces morbidity while achieving superior cosmetic outcomes. Among various sclerosing agents, Bleomycin has gained popularity due to its mechanism of disrupting cellular functions in the abnormal lymphatic endothelial cells, leading to regression of the lesion.

Since its introduction to Vietnam in 2016, Bleomycin has been increasingly used as an adjunctive therapy for lymphangiomas. Despite its growing clinical application, there is a significant lack of comprehensive studies evaluating the safety, efficacy, and long-term outcomes of Bleomycin sclerotherapy in treating pediatric lymphatic malformations, particularly in the Vietnamese population. To date, no large-scale studies have assessed the clinical impact and quality-of-life outcomes of Bleomycin treatment for LM in children within the Vietnamese context. This study seeks to fill this gap in knowledge by comprehensively evaluating the long-term outcomes of intralesional Bleomycin injections in pediatric patients with lymphatic malformations treated at the National Children's Hospital in Vietnam.

The primary objective of this study is to evaluate the safety, efficacy, and long-term outcomes of intralesional Bleomycin injection for pediatric patients diagnosed with lymphatic malformations. The research will focus on both clinical success (such as reduction in lesion size and recurrence rates) and the cosmetic and health-related quality of life (QoL) improvements observed in the patients post-treatment. The study will also examine whether Bleomycin can effectively reduce the need for additional surgical interventions, thus improving both functional and aesthetic outcomes for these children.

This retrospective study will involve a cohort of more than 800 pediatric patients diagnosed with lymphatic malformations and treated with Bleomycin injections at the National Children's Hospital between 2018 and 2022. These patients will be evaluated for safety and efficacy by reviewing their medical records, monitoring for complications, and assessing the recurrence rates of lymphangiomas after treatment. Additionally, long-term cosmetic outcomes will be evaluated using validated patient-reported measures, such as the Patient Scar Assessment Questionnaire (PSAQ), and health-related quality of life will be assessed using the Short Form-36 (SF-36) health survey.

The study aims to assess the safety and efficacy of Bleomycin injection in pediatric patients diagnosed with lymphatic malformations at the National Children's Hospital between 2018 and 2022. This will be done by focusing on post-treatment complications and recurrence rates. Furthermore, the research intends to evaluate the long-term clinical outcomes, including lesion regression, recurrence, and the need for additional interventions. This will help assess the impact of Bleomycin on lesion size, post-treatment complication rates, and the overall clinical success of the intervention.

Another important goal of the study is to analyze the cosmetic outcomes and health-related quality of life in pediatric patients treated with Bleomycin sclerotherapy. The study will use standardized assessment tools like the PSAQ for scarring and the SF-36 for overall health outcomes. These tools will help quantify the patient-reported perception of treatment effects, including both cosmetic outcomes (scar appearance and symptoms) and overall well-being.

Additionally, the study will investigate the role of Bleomycin as a standalone treatment or in combination with surgical interventions to enhance treatment success while minimizing risks and complications associated with invasive procedures. By comparing these approaches, the research aims to determine if Bleomycin alone is sufficient or if a multimodal approach is more effective in treating lymphangiomas.

The results of this study will provide important insights into the feasibility and effectiveness of Bleomycin as an alternative to traditional surgical excision for the treatment of pediatric lymphangiomas. By examining both objective clinical outcomes and subjective patient-reported outcomes, such as quality of life and scar perception, this research will offer a comprehensive understanding of the benefits and challenges of using Bleomycin for this indication. The findings are expected to influence the clinical management of lymphangiomas in pediatric patients, offering evidence-based recommendations on the use of Bleomycin as a safe, effective, and cosmetically favorable treatment option.

Additionally, the study will contribute to filling the gap in local research on the use of Bleomycin for lymphatic malformations in Vietnam, a country where the clinical application of this agent has been relatively new and unstudied. The results of this research could lead to the establishment of evidence-based guidelines for Bleomycin treatment in the Vietnamese healthcare system, supporting its wider adoption as a standard therapy for lymphangiomas.

The study will be conducted with a strict ethical framework, ensuring that all patients and their families provide informed consent before participation, and that their privacy and confidentiality are strictly maintained. Data will be anonymized and stored securely throughout the research process. The findings will be disseminated through peer-reviewed scientific journals, with a particular focus on journals related to pediatric surgery, dermatology, and vascular anomalies, which could help raise awareness of Bleomycin's potential as a viable therapeutic option in the management of lymphangiomas.

In conclusion, this study will not only provide critical clinical data on the efficacy and safety of Bleomycin for treating pediatric lymphangiomas, but it will also enhance our understanding of the long-term cosmetic outcomes and quality of life improvements associated with this treatment. By offering a minimally invasive, less risky alternative to surgical excision, Bleomycin could revolutionize the management of lymphatic malformations in children, improving their health outcomes and overall well-being while minimizing the physical and psychological impact of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age: Pediatric patients under the age of 18 years.
* Diagnosis: Confirmed diagnosis of lymphangioma (lymphatic malformation).
* Location of Lesions: Lymphangiomas located in the head and neck, axilla, abdomen, thorax, groin, or extremities.
* Treatment History: No prior treatment with Bleomycin for lymphangioma.
* Health Status: No serious comorbidities or medical conditions that could interfere with the study or treatment process.
* Informed Consent: Patients (or their legal guardians) provide informed consent to participate in the study.

Exclusion Criteria:

* Age: Patients over the age of 18 years.
* Pregnancy: Pregnant or breastfeeding patients.
* Other Treatments: Patients who have received prior treatments with Bleomycin for lymphangioma.
* Severe Comorbidities: Presence of serious comorbidities (e.g., uncontrolled cardiovascular disease, active infections) that may interfere with the study or treatment process.
* Allergy: Known allergy or hypersensitivity to Bleomycin or any of its components.
* Active Infections: Patients with active local or systemic infections at the time of enrollment.
* Immunosuppression: Immunocompromised patients (due to illness or medications).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of pediatric patients for this study will consist of children under the age of 18 who have been diagnosed with lymphangiomas (lymphatic malformations). These patients will have a variety of lesion locations, including the head and neck, axilla (armpit), abdomen, thorax (chest), groin, or extremities. The age range will encompass infants, children, and adolescents. They might or might not have received previous treatment with Bleomycin or other interventions for lymphatic malformations. Additionally, they might or might not serious comorbidities such as uncontrolled systemic diseases or immunosuppressive conditions. The cohort will be selected from the patient population at the National Children's Hospital, and participants will be enrolled based on a confirmed diagnosis of lymphangioma from 2018 to 2022.
Sampling Method: Non-Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Change in Lesion Size | Through study completion, an average of 5 years
  The degree of lesion size change will be measured to assess the efficacy of intralesional Bleomycin injection. This will be evaluated through clinical examination and imaging techniques (e.g., ultrasound or MRI) to determine the extent of regression of the lymphangioma.
Recurrence Rate | Through study completion, an average of 5 years
  This outcome will track the recurrence rate of lymphangiomas after treatment with Bleomycin. Recurrence is defined as the reappearance or regrowth of the lesion after an initial reduction in size following treatment.
Adverse Reactions | 1 week after each injection
  The safety of the Bleomycin treatment will be assessed by monitoring adverse reactions, including infection, bleeding, swelling, or allergic reactions at the injection site, as well as any systemic side effects.
Number of Injections Required for Remission | Through study completion, an average of 5 years
  The number of Bleomycin injections required to achieve remission (defined as significant size reduction or complete resolution of the lesion) will be recorded. This will help assess the treatment protocol's efficiency and the typical treatment burden for patients.
Proportion of patients requiring additional interventions | Through study completion, an average of 5 years
  This outcome will track the proportion of patients requiring additional interventions (e.g., surgical excision or further sclerotherapy sessions) after the initial Bleomycin treatment. The goal is to determine if Bleomycin alone is sufficient to treat the lymphangiomas or if supplementary interventions are necessary.
PSAQ score - Cosmetic Outcomes and Scar Perception | Through study completion, an average of 5 years
  Cosmetic outcomes and patient scar perception were evaluated using the Patient Scar Assessment Questionnaire (PSAQ). This validated tool includes multiple subscales assessing appearance, symptoms, consciousness, and satisfaction with appearance. Each subscale is scored on a 4-point Likert scale, with individual item scores ranging from 1 to 4, where lower scores indicate better cosmetic outcomes and greater patient satisfaction. The minimum total score is 18, and the maximum is 72, with lower total scores representing more favorable scar outcomes.
SF-36 score - Health-Related Quality of Life (QoL) | Through study completion, an average of 5 years
  Health-related quality of life was assessed using the Short Form-36 Health Survey (SF-36), a validated instrument comprising 36 items across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health perceptions. Scores for each domain range from 0 to 100, with higher scores indicating better health-related quality of life. Both individual domain scores and composite physical and mental component summary scores were analyzed.

SECONDARY OUTCOMES:
Follow-Up Time | Through study completion, an average of 5 years
  The duration of follow-up visits post-treatment will be tracked to monitor for recurrence or complications. Follow-up time will also help assess the long-term effectiveness of Bleomycin treatment.
Time to Regrowth of Lesion | Through study completion, an average of 5 years
  This outcome will measure the time to regrowth of the lymphangioma lesion after initial Bleomycin treatment. The time period between treatment and the first signs of regrowth will be monitored to evaluate the durability of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Quang T Nguyen, M.D., Principal Investigator — Department of Pediatric Surgery, The National Hospital of Pediatrics, Hanoi, Vietnam
Locations (1):
- Department of Surgery, The National Children Hospital, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porwal PK, Dubey KP, Morey A, Singh H, Pooja S, Bose A. Bleomycin Sclerotherapy in Lymphangiomas of Head and Neck: Prospective Study of 8 Cases. Indian J Otolaryngol Head Neck Surg. 2018 Mar;70(1):145-148. doi: 10.1007/s12070-017-1243-x. Epub 2018 Jan 8. PMID 29456959
- [Background] Ameh EA, Nmadu PT. Cervical cystic hygroma: pre-, intra-, and post-operative morbidity and mortality in Zaria, Nigeria. Pediatr Surg Int. 2001 Jul;17(5-6):342-3. doi: 10.1007/s003830000558. PMID 11527161
- [Background] Acevedo JL, Shah RK, Brietzke SE. Nonsurgical therapies for lymphangiomas: a systematic review. Otolaryngol Head Neck Surg. 2008 Apr;138(4):418-24. doi: 10.1016/j.otohns.2007.11.018. PMID 18359347
- [Background] Bawazir OA, Bawazir R, Bawazir A, Kausar N, Said H. Efficacy and Clinical Outcomes of Bleomycin in the Treatment of Lymphangiomas: A Multicenter Experience. Dermatol Surg. 2021 Jul 1;47(7):948-952. doi: 10.1097/DSS.0000000000002976. PMID 33625132
- [Background] Yang Y, Sun M, Ma Q, Cheng X, Ao J, Tian L, Wang L, Lei D. Bleomycin A5 sclerotherapy for cervicofacial lymphatic malformations. J Vasc Surg. 2011 Jan;53(1):150-5. doi: 10.1016/j.jvs.2010.07.019. Epub 2010 Sep 16. PMID 20843632
- [Background] Parashar G, Shankar G, Sahadev R, Santhanakrishnan R. Intralesional Sclerotherapy with Bleomycin in Lymphatic Malformation of Tongue an Institutional Experience and Outcomes. J Indian Assoc Pediatr Surg. 2020 Mar-Apr;25(2):80-84. doi: 10.4103/jiaps.JIAPS_2_19. Epub 2020 Jan 28. PMID 32139985
- [Background] Durani P, McGrouther DA, Ferguson MW. The Patient Scar Assessment Questionnaire: a reliable and valid patient-reported outcomes measure for linear scars. Plast Reconstr Surg. 2009 May;123(5):1481-1489. doi: 10.1097/PRS.0b013e3181a205de. PMID 19407619
- [Background] Contopoulos-Ioannidis DG, Karvouni A, Kouri I, Ioannidis JP. Reporting and interpretation of SF-36 outcomes in randomised trials: systematic review. BMJ. 2009 Jan 12;338:a3006. doi: 10.1136/bmj.a3006. PMID 19139138
- [Background] Ardicli B, Karnak I, Ciftci AO, Tanyel FC, Senocak ME. Sclerotherapy with bleomycin versus surgical excision for extracervical cystic lymphatic malformations in children. Surg Today. 2016 Jan;46(1):97-101. doi: 10.1007/s00595-015-1128-0. Epub 2015 Feb 15. PMID 25682445
- [Background] Upadhyaya VD, Bhatnagar A, Kumar B, Neyaz Z, Kishore JS, Sthapak E. Is multiple session of intralesional bleomycin mandatory for complete resolution of macrocystic lymphatic malformation? Indian J Plast Surg. 2018 Jan-Apr;51(1):60-65. doi: 10.4103/ijps.IJPS_154_17. PMID 29928081
- [Background] Baskin D, Tander B, Bankaoglu M. Local bleomycin injection in the treatment of lymphangioma. Eur J Pediatr Surg. 2005 Dec;15(6):383-6. doi: 10.1055/s-2005-872922. PMID 16418953
- [Background] Wassef M, Blei F, Adams D, Alomari A, Baselga E, Berenstein A, Burrows P, Frieden IJ, Garzon MC, Lopez-Gutierrez JC, Lord DJ, Mitchel S, Powell J, Prendiville J, Vikkula M; ISSVA Board and Scientific Committee. Vascular Anomalies Classification: Recommendations From the International Society for the Study of Vascular Anomalies. Pediatrics. 2015 Jul;136(1):e203-14. doi: 10.1542/peds.2014-3673. Epub 2015 Jun 8. PMID 26055853
- [Background] Tiwari P, Pandey V, Bera RN, Sharma SP, Chauhan N. Bleomycin sclerotherapy in lymphangiomas of the head and neck region: a prospective study. Int J Oral Maxillofac Surg. 2021 May;50(5):619-626. doi: 10.1016/j.ijom.2020.09.008. Epub 2020 Oct 12. PMID 33059994